CLINICAL TRIAL: NCT03510728
Title: Efficacy and Mechanisms of Technology-based Behavioral Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: James M. Henson (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, James M. Henson, Associate Professor of Psychology, Old Dominion University
Organization: Old Dominion University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: OldDominionU; 5R01AA023197 (NIH)
Record Dates: First submitted 2018-04-16; First posted 2018-04-27 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: College Student Drinking
Keywords: Protective Behavioral Strategies
MeSH Terms: conditions — Alcohol Drinking in College

STUDY DESIGN:
Intervention Model Description: There are three conditions at the start of the study regarding assignment to a single-session intervention: none (control), standard BMI (CDCU), and the standard BMI plus a PBS-component. These are crossed with the type of application for their phone: an ecological momentary assessment-only or an ecological momentary intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- No single-session intervention-EMA (No Intervention): Participants will be assessed both using a computer and using their phone. However, they will not receive an intervention at the start of the study and will only be using their phone for ecological assessment only data collection.
- Standard single-session intervention-EMA (Active Comparator): Participants will take a computerized BMI with known efficacy, the college drinker's check up, and will be followed up. Participants in this condition will interact with their phone only for assessment purposes.
  Interventions: Behavioral: college drinker's check up
- Augment single-session intervention-EMA (Experimental): Participants will take a computerized BMI with known efficacy, the college drinker's check up, and will also take a computerized intervention developed to increase the use of protective behavioral strategies during drinking (Protective Behavioral Strategies Intervention). Participants in this condition will interact with their phone only for assessment purposes.
  Interventions: Behavioral: college drinker's check up; Behavioral: Protective Behavioral Strategies Intervention
- No single-session intervention-EMI (Experimental): Participants in this group will not take a single-session intervention at baseline, but will be interacting with their phones during drinking occasions to promote protective behavioral strategy use (Ecological Momentary Intervention).
  Interventions: Behavioral: Ecological Momentary Intervention
- Standard single-session intervention-EMI (Experimental): Participants will take a computerized BMI with known efficacy, the college drinker's check up, and will be followed up. Participants in this condition will be interacting with their phones during drinking occasions to promote protective behavioral strategy use (Ecological Momentary Intervention).
  Interventions: Behavioral: college drinker's check up; Behavioral: Ecological Momentary Intervention
- Augment single-session intervention-EMI (Experimental): Participants will take a computerized BMI with known efficacy, the college drinker's check up, and will also take a computerized intervention developed to increase the use of protective behavioral strategies during drinking (Protective Behavioral Strategies Intervention). Participants in this condition will be interacting with their phones during drinking occasions to promote protective behavioral strategy use (Ecological Momentary Intervention).
  Interventions: Behavioral: college drinker's check up; Behavioral: Protective Behavioral Strategies Intervention; Behavioral: Ecological Momentary Intervention

INTERVENTIONS:
Behavioral: college drinker's check up — The College Drinker's Check-up (CDCU) is a single session, computer-based brief motivational intervention for heavy drinking college students. It takes a student about 45 minutes to go through it.
  Arms: Augment single-session intervention-EMA; Augment single-session intervention-EMI; Standard single-session intervention-EMA; Standard single-session intervention-EMI
Behavioral: Protective Behavioral Strategies Intervention — This intervention component focuses on educating and promoting PBS activities in future college drinking situations
  Arms: Augment single-session intervention-EMA; Augment single-session intervention-EMI
Behavioral: Ecological Momentary Intervention — This EMI is delivered during drinking situations and focuses on promoting PBS use during that particular drinking situation.
  Arms: Augment single-session intervention-EMI; No single-session intervention-EMI; Standard single-session intervention-EMI

SUMMARY:
Large scale surveys indicate that approximately 68% of college students drink alcohol every month and 40% of college students engage in heavy episodic drinking. Despite prevention/intervention efforts, problematic alcohol consumption among college students continues to result in an estimated 1,800 deaths and 600,000 injuries annually, and epidemiological studies demonstrate no appreciable decrease in risk among college students. The purpose of the proposed research is to improve extant college-drinking interventions by advancing the dissemination methodology and the intervention content (Specific Aim 1). As a methodological improvement, rapid advances in mobile computing makes ecological momentary interventions (EMIs) increasingly feasible. EMIs refer to interventions that can be delivered multiple times and "in the moment". EMIs can optimize the timing and location of the intervention while also increasing the dose of the intervention. To improve the intervention content, the researchers will examine protective behavioral strategies (PBS) to reduce alcohol problems, not just alcohol use. PBS are behaviors that one can engage in immediately prior to, during, and immediately following alcohol use that limit alcohol use and/or alcohol-related harm. Research suggests that PBS use can protect individuals from alcohol problems above and beyond its effect on reducing alcohol use. The primary purpose of this research is to provide a more powerful test of a PBS intervention's effects on alcohol-related consequences by using a technology-based intervention methodology (i.e., EMI). Participants will be randomized into to a fully crossed, 3 (Standard BMI, BMI with a PBS component, control) X 2 (PBS-based EMI, Ecological Assessment Only) design. These 6 conditions will answer several critically important research questions (Specific Aim 2): a) does the addition of a PBS component improve the efficacy of a standard BMI, b) does a PBS-based EMI improve efficacy over the standard, single session BMI, c) does the combination of motivation-based intervention (BMI) with a skills-based intervention (EMI) yield even greater decreases in consequences (i.e., moderation). A final purpose of this research is to examine PBS norms, PBS perceived effectiveness, and motivation to change PBS use as novel mediators of the improved interventions. Results can be used to disseminate more effective college drinking interventions that are cheaper and more efficacious.

DETAILED DESCRIPTION:
Hazardous alcohol use among college students is a significant public health concern that has resulted in the development of numerous interventions. Although motivational interviewing components are effective at reducing problematic alcohol consumption among college students via reductions in descriptive norms (i.e., the perceived drinking by peers), the effects of single-session brief motivational interventions (BMIs) on alcohol use and consequences are relatively short-lived (i.e., 3 months). Guided by a harm-reduction perspective, researchers have become increasingly interested in how protective behavioral strategies (PBS) can impact alcohol consequences beyond the effects of reduced alcohol consumption. PBS have been found to be a robust predictor of alcohol-related problems controlling for consumption, and multiple intervention studies have found that PBS mediates intervention effects. Few studies, however, have examined the efficacy of PBS-related intervention components.

Specific Aim 1a: The researchers will augment and improve extant college alcohol interventions by developing and rigorously evaluating an added PBS component to an existing BMI with demonstrated efficacy to further reduce alcohol-related consequences beyond what is explained by reduced consumption.

An additional goal of this research is to deliver PBS in a way that capitalizes on newer technologies that allow for the repeated in vivo delivery of alcohol interventions. Given the widespread use of handheld devices among the college population, ecological momentary intervention (EMI) shows great promise in producing lasting behavior for a modest cost.

Specific Aim 1b: The researchers will develop a technology-based, college-drinking ecological momentary intervention (EMI; a newer, less explored methodology) that is disseminated using mobile, hand-held devices, which can be used in vivo with every drinking episode.

Characterizing Intervention Efficacy. The researchers intend to demonstrate that adding a PBS-focused component can increase efficacy beyond standard single-session BMIs while keeping costs minimal. Although the researchers predict that the PBS-based EMI will effect greater and more lasting decreases in alcohol consequences beyond standard intervention, it is important to verify that cheaper, single-session alternatives are not as effective (i.e., PBS-based BMI). Therefore, the researchers intend to implement a 2 (EMI, Ecological Momentary Assessment only [EMA]) by 3 (no single-session intervention control, standard BMI, BMI plus PBS component) factorial design. The researchers will characterize the efficacy of the BMI+PBS and EMI over traditional, single-session BMIs in several ways:

Specific Aim 2a: The researchers will examine whether the EMI methodology effects greater and more lasting behavior change as compared to the EMA assessment conditions.

To accomplish Specific Aim 2a, the researchers will examine the main effect of assessment (EMI vs. EMA) to demonstrate that the EMI conditions yield better longitudinal outcomes regardless of the single-session intervention.

Specific Aim 2b: The researchers will examine whether the PBS intervention component leads to reduced alcohol related consequences as compared to a standard BMI, even with a single-session intervention.

To accomplish Specific Aim 2b, the researchers will examine the main effect of the single-session intervention to demonstrate that a single-session BMI that has been enhanced by the PBS component will yield superior longitudinal effects relative to a BMI without the PBS component regardless of assessment style (EMA or EMI); the researchers further expect both BMI groups to be superior to the no-intervention control.

Specific Aim 2c: The researchers expect the EMI to moderate the single-session intervention, such that the PBS-BMI coupled with EMI will yield superior longitudinal outcomes on drinking consequences.

The researchers expect the PBS intervention component to be most efficacious when delivered in vivo during high-risk, alcohol use situations (i.e., EMI), where student motivation and perceived norms about drinking are most challenged. By using a 2X3 design, the researchers will be able to verify the synergistic interaction and characterize the effect size of the relative superiority of the PBS single-session component coupled with the PBS-based EMI.

Mechanisms of Behavior Change. Unlike the BMI, which relies upon motivation and descriptive norm changes, the researchers expect the PBS intervention component to have different mechanisms of behavior change. Specifically, the PBS component is an intervention that emphasizes skill use rather than motivation. Further, when coupled with EMI, which is a direct behavioral intervention, the PBS component will effect change by targeting specific behaviors as opposed to drinking motivation.

Specific Aim 3: To characterize the differential mechanisms of behavior change across the single-session and EMI interventions.

The researchers expect key differences in the mediating variables across interventions conditions. The researchers will examine PBS norms, PBS perceived effectiveness, and motivation to change PBS to ascertain how the researchers can best effect increases in PBS use in college populations.

ELIGIBILITY:
Inclusion Criteria:

* Current college students at the sponsor institution at the time of enrollment
* Between the ages of 18 and 25
* Consumed at least standard drink of alcohol in the past 4 weeks

Exclusion Criteria:

* Under age of 18 or older than 25
* Not a college student
* Did not drink alcohol in the past 4 weeks

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Alcohol Consumption | 6-months
  Alcohol Use Disorders Identification Test (general consumption)
Alcohol Consumption | 6-months
  Modified version of the Daily Drinking Questionnaire (typical weekly consumption)

SECONDARY OUTCOMES:
Alcohol Consequences | 6-months
  Young Adult Alcohol Consequences Questionnaire

OTHER OUTCOMES:
Mechanisms of behavior change (PBS use) | 6-months
  Revised Protective Behavioral Strategies Scale is used to measure the use of three types of protective behavioral strategies: Manner of Drinking, Limiting/Stopping Drinking, and Serious Harm Reduction. Each scale is averaged (possible range 1 - 6, 1 = not at all, 6 = always/almost always), higher scores indicate more use of protective behavioral strategies.
Mechanisms of behavior change (PBS helpfulness) | 6-months
  Perceived PBS Helpfulness scale assess the perceived helpfulness of using various PBS behaviors to moderate drinking. Items are assessed on a 1 (Not helpful) to 5 (Extremely helpful) scale.
Mechanisms of behavior change (PBS motivation) | 6-months
  The Motivation to use PBS scale assess the motivation of using various PBS behaviors to moderate drinking. Items are assessed on a 1 (Not motivated) to 5 (Extremely motivated) scale.
Mechanisms of behavior change (PBS intentions) | 6-months
  The Intentions to use PBS scale assess the future intentions of using various PBS behaviors to moderate drinking. Items are assessed on a 1 (Never) to 5 (Always) scale.

CONTACTS AND LOCATIONS:
Overall Officials: James M Henson, Ph.D., Principal Investigator — Old Dominion University
Locations (5):
- United States (5):
  - California State University Dominguez Hills, Carson, California
  - Colorado State University, Fort Collins, Colorado
  - University of New Mexico, Albuquerque, New Mexico
  - Old Dominion University, Norfolk, Virginia
  - William and Mary, Williamsburg, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Collins RL, Parks GA, Marlatt GA. Social determinants of alcohol consumption: the effects of social interaction and model status on the self-administration of alcohol. J Consult Clin Psychol. 1985 Apr;53(2):189-200. doi: 10.1037//0022-006x.53.2.189. No abstract available. PMID 3998247
- [Background] Read JP, Kahler CW, Strong DR, Colder CR. Development and preliminary validation of the young adult alcohol consequences questionnaire. J Stud Alcohol. 2006 Jan;67(1):169-77. doi: 10.15288/jsa.2006.67.169. PMID 16536141
- [Background] Martens MP, Ferrier AG, Sheehy MJ, Corbett K, Anderson DA, Simmons A. Development of the Protective Behavioral Strategies Survey. J Stud Alcohol. 2005 Sep;66(5):698-705. doi: 10.15288/jsa.2005.66.698. PMID 16329461